CLINICAL TRIAL: NCT02945787
Title: Expanding the Reach of a Validated Smoking-Cessation Intervention: A Spanish-Language Trial
Brief Title: Spanish-Language Smoking Cessation Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-18633; R01CA199143 (NIH)
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Smoking Cessation
Keywords: Spanish speaking; self-help; tobacco abstinence; public health; Forever Free; Stop Smoking for Good
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended Self-help (Experimental): Spanish-Language Version of the Stop Smoking for Good: The Extended Self-help condition will comprise the 11 Stop Smoking for Good booklets and 9 supportive My Story pamphlets transcreated for Spanish speaking smokers.
  Interventions: Behavioral: Spanish-Language Version of the Stop Smoking for Good
- Usual Care (UC) (Active Comparator): NCI-Produced Spanish-language Self-help Booklet: The UC control condition enhances the external validity of the study by providing a comparison to an existing, credible intervention that a smoker could receive in a medical setting or elsewhere.
  Interventions: Behavioral: NCI-Produced Spanish-language Self-help Booklet

INTERVENTIONS:
Behavioral: Spanish-Language Version of the Stop Smoking for Good — Participants in the first arm will receive the Spanish-language version of the Stop Smoking for Good (SS-SP) intervention distributed over 18 months.
  Arms: Extended Self-help
Behavioral: NCI-Produced Spanish-language Self-help Booklet — Participants in the second arm will receive a single, credible, NCI-produced Spanish-language self-help booklet.
  Arms: Usual Care (UC)

SUMMARY:
Results of a recently completed National Cancer Institute (NCI) funded trial of an intervention, Forever Free: Stop Smoking for Good, revealed high efficacy throughout the 24- month follow-up period, further supporting the utility of extended self-help for promoting and maintaining tobacco abstinence. Investigators have recognized that wide-scale implementation, and therefore public health impact, would be enhanced by the availability of a Spanish-language version to reach the largest and fastest growing ethnic minority population of smokers.

The goal of this study is to address this gap by testing a Spanish-language version of the validated self-help smoking cessation intervention. If demonstrated effective, the proposed intervention would represent an easily disseminable and low-cost intervention with significant public health impact for Hispanic/Latino smokers throughout the United States. The aims of this project are to test the efficacy of a Spanish-language version of a validated, extended self-help intervention for smoking cessation among Spanish-speaking smokers against usual care control. Participants (N = 1400) recruited nationally will be randomized to the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Smoking ≥ 5 tobacco cigarettes/week over the past year
* Not currently enrolled in a face-to-face smoking cessation program
* Monolingual Spanish-speaking, or bilingual Spanish-English and prefer receiving educational health materials in Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1417 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brandon, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Simmons VN, Sutton SK, Medina-Ramirez P, Martinez U, Brandon KO, Byrne MM, Meade CD, Meltzer LR, Brandon TH. Self-help smoking cessation intervention for Spanish-speaking Hispanics/Latinxs in the United States: A randomized controlled trial. Cancer. 2022 Mar 1;128(5):984-994. doi: 10.1002/cncr.33986. Epub 2021 Oct 22. PMID 34679188
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care (UC): NCI-Produced Spanish-language Self-help Booklet: The UC control condition enhances the external validity of the study by providing a comparison to an existing, credible intervention that a smoker could receive in a medical setting or elsewhere.
  NCI-Produced Spanish-language Self-help Booklet: Participants in the second arm will receive a single, credible, NCI-produced Spanish-language self-help booklet. Outcomes will be assessed through 24 months.
Period: Overall Study
Arm/Group | Extended Self-help | Usual Care (UC)
Started | 714 | 703
Completed | 714 | 703
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Self-help | Usual Care (UC) | Total
Number analyzed (Participants) | 714 | 703 | 1417
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 648 | 643 | 1291
  >=65 years | 66 | 60 | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 346 | 339 | 685
  Male | 368 | 364 | 732
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 30 | 42
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 17 | 13 | 30
  Black or African American | 23 | 18 | 41
  White | 347 | 313 | 660
  More than one race | 20 | 28 | 48
  Unknown or Not Reported | 293 | 301 | 594
Region of Enrollment [Number; unit: participants]
  United States | 714 | 703 | 1417

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Tobacco Abstinence at 6 Months
Description: Participants will complete follow-up assessment packets at 6 month intervals through 24 months. At each assessment point, investigators will calculate 7-day point- prevalence abstinence rates.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Extended Self-help | Usual Care (UC)
Number analyzed (Participants) | 714 | 703
percentage of participants | 21.7 | 11.3

2. Primary Outcome: Percentage of Participants With Tobacco Abstinence at 12 Months
Description: as for outcome 1
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Extended Self-help | Usual Care (UC)
Number analyzed (Participants) | 714 | 703
percentage of participants | 28.4 | 17.0

3. Primary Outcome: Percentage of Participants With Tobacco Abstinence at 18 Months
Description: as for outcome 1
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Extended Self-help | Usual Care (UC)
Number analyzed (Participants) | 714 | 703
percentage of participants | 29.3 | 20.7

4. Primary Outcome: Percentage of Participants With Tobacco Abstinence at 24 Months
Description: as for outcome 1
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Extended Self-help | Usual Care (UC)
Number analyzed (Participants) | 714 | 703
percentage of participants | 33.1 | 23.3

ADVERSE EVENTS:
Time Frame: Adverse events were not collected
Description: Adverse events were not collected
Arm/Group | Extended Self-help | Usual Care (UC)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT02945787/Prot_SAP_000.pdf